CLINICAL TRIAL: NCT04863157
Title: A Sleep Intervention for Children After Cancer: Survivor Sleep Health Information Program (Survivor-SHIP)
Brief Title: Survivor-Sleep Health Information Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Children's Cancer Research Fund (Other)
Responsible Party: Principal Investigator, Eric Zhou, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-018
Record Dates: First submitted 2021-04-21; First posted 2021-04-28 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Sleep Problem; Insomnia; Pediatric Cancer
Keywords: Sleep Problem; Insomnia; Pediatric Cancer; Behavioral Intervention
MeSH Terms: conditions — Parasomnias; Sleep Initiation and Maintenance Disorders; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Survivor-SHIP (Experimental): Parents/guardians will take part in 3 education sessions over a one month period. During the sessions, they will learn more about common sleep problems following cancer treatment and ways to understand their child's unique patterns. They will then be educated about behavioral changes they can make to improve their child's sleep.
  Interventions: Behavioral: Survivor-SHIP

INTERVENTIONS:
Behavioral: Survivor-SHIP — Parent/guardian education about healthy sleep practices to improve their child's sleep health.
  Other Names: Survivor-Sleep Health Information Program

SUMMARY:
The purpose of the study is to learn if an educational program delivered to parents/guardians can help improve the sleep of children experiencing sleep problems after completing cancer treatment. The name of the intervention is Survivor-SHIP (Sleep Health Information Program).

DETAILED DESCRIPTION:
This study will evaluate Survivor-SHIP in a single-arm trial of 20 off-treatment childhood cancer survivors (ages 5-12). The intervention is an adapted version of the family-centered Sleep Health Program designed at Seattle Children's Hospital. The program offers parents information about how to utilize evidence-based strategies for their child's sleep, and has demonstrated success in a community-based sample of children with behavioral sleep problems. Sessions will focus on providing parents with education about healthy sleep and setting targets for modifiable behaviors that can improve their child's sleep health.

The study will include 3 education sessions taking place over videoconference. Families will be asked to track their child's sleep using sleep diaries during the course of the program. Prior to, and following the program, families will be asked to complete study questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 5-12 years, with a history of a cancer diagnosis (except non-melanoma skin cancer).
* No cancer therapy (excluding chemoprevention) in the past 6 months, and no further therapy planned.
* Child meets diagnostic criteria for insomnia disorder as determined by insomnia screening criteria (see Appendix A)
* Parent/guardian is able to read and write in English.
* Regular access to a computer/smartphone with internet access at home.

Exclusion Criteria:

* Reports child has been diagnosed with a Seizure Disorder or has experienced a seizure in the past 12 months.
* Reports child has been diagnosed with a developmental disorder such as Autism Spectrum Disorder, Cerebral Palsy, Fragile X Syndrome, or Moderate to Profound Intellectual Disability.
* Reports child has been diagnosed with sleep apnea, and are not receiving recommended medical treatment for their sleep apnea.
* Intention to adjust (decrease or increase) child's use of any prescribed or over-the-counter sleep medications during the study period.
* Any impairment (e.g., hearing, visual, cognitive) that interferes with the parent/guardian's ability to complete all study procedures independently.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Intervention acceptability | 6 weeks
  Intervention acceptability will be assessed using the Satisfaction subscale of the Usability, Satisfaction, and Ease of use (USE) scale. Total scores will range from 0-11, with higher scores indicating better acceptability.
Intervention feasibility | 6 weeks
  Intervention feasibility will be assessed based on adherence rates to the intervention sessions.

SECONDARY OUTCOMES:
Sleep knowledge | 6 weeks
  The Parent Sleep Knowledge questionnaire is a 10-item questionnaire assessing the parents' knowledge about children's sleep. The scale is scored from 0 to 10, with a higher score indicating more knowledge.
Sleep habits | 6 weeks
  The Children's Sleep Habits Questionnaire (CSHQ) is a 33-item questionnaire that will assess the child's overall sleep habits. A Total Sleep Disturbances score is calculated as the sum of all scored questions, and can range from 33 to 99, with higher scores indicating more sleep disturbance.
Sleep quality | 6 weeks
  The Patient-reported outcomes measurement information system (PROMIS) pediatric sleep scales are an 8-item measure that assesses the child's sleep quality. A total score will range from 8 to 40, with higher scale scores indicating poorer sleep health
General quality of life | 6 weeks
  The child's quality of life will be evaluated by the Pediatric Quality of Life Inventory (PedsQL), a 23-item scale measuring core physical, mental, and social health dimensions. Scores are transformed on a scale from 0 to 100, with higher scores indicating better function.
Screen time | 6 weeks
  The extent of the child's electronic screen use will be assessed by a set of 9 questions that were developed specifically for this study by the Principal Investigator. They assess the duration of electronics usage across different devices and timing of usage.
Sleep change | 6 weeks
  The investigators will assess whether the family implemented any non-intervention advised changes to their child's sleep routine, such as increasing medication for their sleep during the intervention period. This set of 5 questions will be assessed only at the post-intervention timepoint.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Zhou, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu